CLINICAL TRIAL: NCT03800082
Title: Development and Usability Testing of a Progressive WebApp for Women With Heart Disease
Acronym: at heart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Monica Parry, Associate Professor and Coordinator, Nurse Practitioner Programs, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 389044
Record Dates: First submitted 2019-01-04; First posted 2019-01-11 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Pain; Cardiac Ischemia; Women; Pain, Chronic
Keywords: Women, Self-Management, Cardiac Pain
MeSH Terms: conditions — Pain; Coronary Artery Disease; Chronic Pain; Angina Pectoris

STUDY DESIGN:
Intervention Model Description: A two group parallel single blind pilot RCT.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind the participants to group allocation due to the specific nature of the intervention; however, a data analyst at the University of Toronto's Faculty of Nursing who is blinded to treatment allocation will conduct the analysis ensuring neutrality of the outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants allocated to the control group will receive the usual care and supports provided to women with cardiac pain, including usual clinic appointments and follow-up.
- Treatment (Experimental): Participants allocated to the treatment group will also learn how to use the progressive WebApp intervention. The intervention will be delivered on restricted password-protected applications that will permit tracking of adherence (number of logins to app and website using Google Analytics). Participants will be encouraged to log-in regularly to the progressive WebApp (via automated alerts) over the 3-month period to complete a Heart and/or Wellness Check. A Chatbot named 'Holly' will assist women with log-in and maintaining health and wellness. Participants will be directed to the PC for technical problems.
  Interventions: Behavioral: at heart (changed from HEARTPA♀N during usability testing)

INTERVENTIONS:
Behavioral: at heart (changed from HEARTPA♀N during usability testing) — An integrated smartphone and web-based intervention (at heart) to provide evidence-informed symptom triage and self-management support to reduce pain and increase health-related quality of life (HRQoL) in women with heart disease. The intervention for participants randomized to the treatment group will consist of regular use of a progressive WebApp that is managed by a Chatbot named 'Holly', in addition to usual care, for a period of 3 months.
  Arms: Treatment

SUMMARY:
The overall goal of this program of research is to develop and systematically evaluate an integrated smartphone and web-based intervention (at heart [formerly called HEARTPA♀N]) to provide evidence-informed symptom triage and self-management support to reduce pain and increase health-related quality of life (HRQoL) in women with heart disease. The investigators will use the individual and family self-management theory, mobile device functionality and the pervasive information architecture of mHealth interventions, and follow the sequential phased approach recommended by the Medical Research Council (MRC) to develop at heart (progressive WebApp). Funding was received from the Canadian Institutes of Health Research to develop the architecture and conduct usability testing (Phase 2, complete) to ensure it is easy to use, efficient and satisfying to operate. In Phase 3 (current proposal), feasibility in terms of implementation (accrual rates, acceptability and level of engagement) and initial estimation of effectiveness outcomes (estimates of magnitude of effect) will be evaluated in a pilot randomized controlled trial (RCT). The Phase 3 pilot study will enable the investigators to refine the prototype, inform the methodology, and calculate the sample size for a larger multi-site RCT (Phase 4, future work).

DETAILED DESCRIPTION:
Phase 3 (Study 3): Pilot Randomized Controlled Trial of the at heart (formerly called HEARTPA♀N) Intervention.

The at heart intervention is the first of its kind; there are no previous trials of the efficacy of such an intervention to decrease pain and improve HRQoL in women with heart disease. The investigators will undertake a process and preliminary effect evaluation of the intervention for women with heart disease, as guided by the MRC framework. The primary objective is to determine the feasibility of implementing an RCT of the intervention. A process evaluation will be conducted to examine: 1) the feasibility of randomization, recruitment and retention, 2) acceptability and barriers to implementing the intervention (including the symptom triage algorithms), and 3) the extent of engagement with the intervention. The investigators will also undertake a preliminary efficacy evaluation of the primary outcomes. Based on the investigator's theorized mechanism of change, they hypothesize that the intervention will reduce pain and improve HRQoL (primary outcomes). The investigators will assess the variability and sensitivity to change for both outcomes. Prior to conducting a full scale RCT of a complex intervention, such as at heart, the MRC recommends that a pilot trial be performed. Results from this pilot trial will inform the success of a future RCT in three ways: 1) help determine sample size calculation for the full-scale trial, 2) test procedures (recruitment, randomization, follow-up), which will make up the design of the full-scale trial, and 3) test feasibility of implementing the intervention, particularly by estimating rates of recruitment and retention. Triage algorithms and self-management interventions will be developed using a strong theoretical framework, informed by needs assessments and a comprehensive integrated mixed methods systematic review, with preliminary acceptability and usability testing by end-users. The investigators anticipate minimal risk to safety but will track adverse events using the Adverse Event Form. Moreover, latest WebApp technologies have been integrated through the use of a Chatbot named 'Holly'.

ELIGIBILITY:
Inclusion Criteria:

* women greater than 18 years of age with obstructive and non-obstructive CAD pain, post PCI/cardiac surgery pain lasting greater than 3 months
* women will be required to speak and read English

Exclusion Criteria:

* severe cognitive impairment assessed using the Six-Item Screener
* major co-morbid medical or psychiatric illness that could preclude their ability to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We will use the PRAXY Gender Questionnaire - Short Form
Enrollment: 98 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility (recruitment, retention, engagement) | 3 months
  A process evaluation will be used to assess the feasibility of the implementation of the intervention. The PC will track any issues or difficulties encountered during trial implementation, such as problems using the app. Engagement will be assessed using Google Analytics, which will track patterns of app and website usage. Engagement with the app diary will be defined as 100% with daily entries for 3 months. Engagement with goal setting will be defined as 100% when 12 goals are identified over the 3-month period. Criteria for implementation success: recruitment rates > 70%, retention > 85%, minimal technical difficulties reported by < 10%, engagement > 80%, and minimal missed responses. Prevalence of refusal, retention, engagement and technical difficulties reported will be calculated with their 95% confidence intervals.
Feasibility (acceptability, satisfaction) | 3 months
  The investigators will also assess acceptability and satisfaction in all participants in the intervention group using a modified Acceptability e-Scale (AES). The modified AES includes 9 items, each with a 5-point Likert response. Higher scores represent better acceptability/satisfaction. Responses are summed and averaged. Criteria for implementation success: AES mean summary score > 4.

SECONDARY OUTCOMES:
Pain (Brief Pain Inventory) | 3 months
  A preliminary efficacy evaluation will also be undertaken focusing on the outcomes of pain. Pain will be measured using the Brief Pain Inventory-Short Form (BPI-SF), which rates pain severity and the degree to which pain interferes with mood, sleep, and other physical activities such as work, social activity and relations with others. We will investigate the variability and sensitivity to change for pain (T2-T1). We will calculate the number of participants who report clinically meaningful decreases in pain, which has been defined for the BPI-SF as a two-point difference in worst pain. Variability will be estimated using the mean/median scores and standard deviation, in each group separately, at pre and post-test.
Health-related quality of life (HRQOL) | 3 months
  A preliminary efficacy evaluation will also be undertaken focusing on the outcomes of HRQOL. HRQOL will be measured using the SF-36v2TM, which contains 36 items and yields a score for each of the 8 domains of health: physical functioning, role limitations due to physical health (role-physical), bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems (role emotional), and mental health. We will investigate the variability and sensitivity to change for HRQOL (T2-T1). Sensitivity to change will be assessed by determining the number of participants who had a clinically meaningful increase in HRQOL: ≥ 15 points in physical functioning, general health and mental health; ≥ 16.7 in role emotional functioning; ≥ 18.5 points in role physical functioning and vitality; ≥ 20 points in bodily pain; and ≥ 25 points in social functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Parry, PhD, Principal Investigator — University of Toronto
Locations (1):
- Monica Parry, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parry M, Dhukai A, Clarke H, Bjornnes AK, Cafazzo JA, Cooper L, Harvey P, Katz J, Lalloo C, Leegaard M, Legare F, Lovas M, McFetridge-Durdle J, McGillion M, Norris C, Parente L, Patterson R, Pilote L, Pink L, Price J, Stinson J, Uddin A, Victor JC, Watt-Watson J, Auld C, Faubert C, Park D, Park M, Rickard B, DeBonis VS. Development and usability testing of HEARTPAfemale symbolN: protocol for a mixed methods strategy to develop an integrated smartphone and web-based intervention for women with cardiac pain. BMJ Open. 2020 Mar 9;10(3):e033092. doi: 10.1136/bmjopen-2019-033092. PMID 32156763